CLINICAL TRIAL: NCT01480453
Title: Retrospective and Prospective Post Market Clinical Follow-up Study of the Zimmer Trabecular Metal Humeral Stem
Brief Title: Outcomes Study of the TM Humeral Stem Used in Primary, Total or Hemi Shoulder Arthroplasty
Status: Terminated | Type: Observational
Why Stopped: Business decision was made to remove the CE mark from this product, thus prompting the closing of this study.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CMU2010-29E
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Post-traumatic Arthritis; Ununited Humeral Head Fracture; Irreducible 3- and 4-part Proximal Humeral Fractures; Avascular Necrosis
Keywords: Osteoarthritis; Rheumatoid arthritis; Post-traumatic arthritis; Ununited humeral head fracture; Irreducible 3- and 4-part proximal humeral fractures; Avascular necrosis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Trabecular Metal Humeral Stem: Patients requiring primary, total or hemi shoulder arthroplasty who receive the Trabecular Metal Humeral Stem.
  Interventions: Device: Trabecular Metal Humeral Stem

INTERVENTIONS:
Device: Trabecular Metal Humeral Stem — Trabecular Metal Humeral Stem used in primary, total or hemi shoulder arthroplasty
  Other Names: TM Humeral Stem; TM Humeral

SUMMARY:
The objectives of this study are to obtain survival and outcome data on the Trabecular Metal Humeral Stem when used in primary, total or hemi shoulder arthroplasty.

DETAILED DESCRIPTION:
The objectives of this study are to obtain survival and outcome data on the Trabecular Metal Humeral Stem when used in primary, total or hemi shoulder arthroplasty. This will be done by analysis of standard scoring systems, radiographs and adverse event records. Data will be collected and analyzed to monitor pain, function, and survivorship and to confirm the performance of the Trabecular Metal Humeral Stem.

Performance will be evaluated by monitoring the frequency and incidence of adverse events as well as by assessment of the overall pain and functional performances, survivorship, health status and radiographic parameters of all enrolled study subjects who receive the Trabecular Metal Humeral Stem.

Pain and functional performance will be measured using the American Shoulder and Elbow Surgeons (ASES) Shoulder Assessment and the Single Assessment Numeric Evaluation (SANE), survivorship will be based on removal or intended removal of the device, health status will be determined by evaluation of the SF-12 as well as AEs and radiographic parameters by analysis of x-rays.

ELIGIBILITY:
Inclusion Criteria:

* Patient is >18 years of age;
* Patient is skeletally mature;
* Patient qualifies for primary unilateral or bilateral total or hemi shoulder arthroplasty based on physical exam and medical history including the following: Osteoarthritis, Rheumatoid arthritis, Post-traumatic arthritis, Ununited humeral head fracture, Irreducible 3- and 4-part proximal humeral fractures, Avascular necrosis
* Patient is willing and able to provide written informed consent;
* Patient is willing and able to cooperate in the required post-operative therapy;
* Patient is will and able to complete scheduled follow-up evaluations/questionnaires as described in the Informed Consent;
* Patient has participated in the Informed Consent process and has signed the IRB/ERB approved informed consent;

Exclusion Criteria:

* The patient is a prisoner;
* The patient is mentally incompetent or unable to understand what participation in the study entails;
* The patient is a known alcohol or drug abuser;
* The patient is anticipated to be non-compliant;
* The patient has one of the following compromising the affected limb; a significant injury to the upper brachial plexus, paralysis of the axillary nerve or a neuromuscular disease compromising the affected limb which would render the procedure unjustifiable;
* The patient has a local/systemic infection;
* The patient is known to be pregnant;
* The patient has marked bone loss;
* The patient has a known sensitivity or allergic reaction to one or more of the implanted materials;
* The patient is unwilling or unable to give consent or to comply with the follow-up program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each investigator will screen from his/her patients who suffer from Osteoarthritis, Rheumatoid arthritis, Post-traumatic arthritis, Ununited humeral head fracture, Irreducible 3- and 4-part proximal humeral fractures, Avascular necrosis who meet the inclusion/exclusion criteria stated in the protocol.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2011-01-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Survivorship | 10 Years
  Based on removal or intended removal of the device and determined using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Pain and Functional Performance | 10 Years
  Measurements will be based on the American Shoulder and Elbow Surgeons (ASES) Shoulder Assessment and the Single Assessment Numeric Evaluation (SANE)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Norton Orthopaedic Specialists, Louisville, Kentucky
  - William Beaumont Hospital, Royal Oak, Michigan
  - The Rothman Institute, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided